CLINICAL TRIAL: NCT01335581
Title: A Study of the RevLite Q-Switched Nd:YAG Laser System With Smart Infinite (SI) Handpiece for the Treatment of Refractory Mixed Type Melasma
Brief Title: Study of Laser Treatment of Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConBio, a Cynosure Company (Industry)
Responsible Party: Sponsor
Organization: Cynosure, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C69-10-M
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Results first posted 2020-12-28 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Refractory Mixed Type Melasma
MeSH Terms: interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser treatment (Experimental): Laser treatment and microdermabrasion and topical lightening agent regimen
  Interventions: Device: Q-Switched Nd:YAG Laser (RevLite); Drug: Retin-A and microdermabrasion
- Control (Active Comparator): Microdermabrasion and topical lightening agent regimen
  Interventions: Drug: Retin-A and microdermabrasion

INTERVENTIONS:
Device: Q-Switched Nd:YAG Laser (RevLite) — Laser treatment added to a microdermabrasion and topical lightening agent regimen
  Arms: Laser treatment
Drug: Retin-A and microdermabrasion — Microdermabrasion and topical lightening agent regimen

SUMMARY:
The purpose of this study is to evaluate the RevLite laser in the treatment of refractory mixed type melasma.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type III-VI
* mixed (epidermal and dermal) melasma diagnosed by Wood's Lamp exam
* age 18 or older
* melasma persisting for greater than 6 months that has failed to respond to conventional treatment with hydroquinone or other topical lightening agents
* written and verbal informed consent
* willing and able to comply with study instructions and return to the clinic for required visits

Exclusion Criteria:

* Pregnancy, breastfeeding, taking birth control pills or plans to become pregnant during the study
* history of cutaneous photosensitization, porphyria, and hypersensitivity to porphyrins or photodermatosis
* any skin pathology or condition that could interfere with the evaluation or requires the use of interfering topical or systemic therapy
* uncorrected coagulation defect or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy)
* any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study
* currently enrolled in an investigational drug or device trial, or has received an investigational drug or has been treated with an investigational device within 30 days prior to entering this study
* inability to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function
* unreliability for the study (this includes subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits)
* use of photosensitizing drugs within a timeframe where photosensitization from these drugs may still be present
* need to be exposed to artificial tanning devices or excessive sunlight during the trial
* Diabetes Type I or II
* sensitivity to hydroquinone or Retin-A
* evidence of a compromised immune system or hepatitis
* use of bleaching creams or retinoids within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Kauvar, MD, Principal Investigator — New York Laser and Skin Care
Locations (1):
- New York Laser and Skin Care, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser Treatment: Laser treatment added to microdermabrasion and topical lightening agent regimen
  Q-Switched Nd:YAG Laser (RevLite): Laser treatment added to a microdermabrasion and topical lightening agent regimen
- Control Group: Microdermabrasion and skin lightening regimen
Period: Overall Study
Arm/Group | Laser Treatment | Control Group
Started | 9 | 9
Completed | 5 | 3
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Microdermabrasion and topical lightening agent regimen
- Total: Total of all reporting groups
Arm/Group | Laser Treatment | Control Group | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 4 | 5 | 9
  Race/Ethnicity: Spanish/Hispanic | 2 | 2 | 4
  Race/Ethnicity: African American | 0 | 2 | 2
  Race/Ethnicity: Indian | 2 | 0 | 2
  Race/Ethnicity: Asian-American | 1 | 0 | 1
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Type I | 0 | 0 | 0
    Fitzpatrick Skin Type II | 0 | 0 | 0
    Fitzpatrick Skin Type III | 3 | 3 | 6
    Fitzpatrick Skin Type IV | 4 | 4 | 8
    Fitzpatrick Skin Type V | 2 | 2 | 4
    Fitzpatrick Skin Type VI | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Melasma Area Severity Assessment (MASI) Score Change From Baseline to Follow Up
Description: The severity of the melasma is assessed based on a photographic scale. The scale ranges from 0 to 48, with 48 being the most severe. A decrease in the MASI score from the baseline to the follow up corresponds with decreasing severity.
Time Frame: 3 Months
Population: 8 subjects did not attend the 3 month follow up, and 2 subjects attended but did not complete their MASI score.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: Lightening cream and microdermabrasion only.
Arm/Group | Laser Treatment | Control Group
Number analyzed (Participants) | 5 | 3
score on a scale | -5.6 (6.9) | 4.7 (9.2)

ADVERSE EVENTS:
Time Frame: Adverse Events occurring were captured and followed throughout each patient's duration in the study, approximately 11 months.
Description: Only 1 subject experienced adverse events during this study.
Groups:
- Control Group: Microdermabrasion and topical lightening agent regimen only.
Arm/Group | Laser Treatment | Control Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Treatment (N=9) | Control Group (N=9)
Dryness (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.